CLINICAL TRIAL: NCT04807699
Title: Rede Colaborativa Para Geração de Evidência Científica em COVID-19 Para o Sistema Único de Saúde no Brasil - RECOVER SUS-BRASIL
Brief Title: Collaborative Network for Generating Scientific Evidence in COVID-19 For the Unified Health System in Brazil - RECOVER SUS-BRASIL
Acronym: Recoversus
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Evandro Chagas National Institute of Infectious Disease (Other)
Collaborators: Hospital Universitario Pedro Ernesto (Other); Universidade Federal do Rio de Janeiro (Other); Hospital Couto Maia/SES/BA (Unknown); Hospital São José de Doenças Infecciosas - HSJ / Secretaria de Saúde Fortaleza (Unknown); Hospital Estadual Sumaré Dr. Leandro Francheschini (Unknown); Universidade Federal de Santa Maria (Other); Hospital Regional de São José - Dr. Homero de Miranda Gomes (Other); Hospital dos Servidores do Estado do Rio de Janeiro (Other Government); Federal University of Minas Gerais (Other); Gaffree & Guinle Universitary Hospital (Other); Hospital Nossa Senhora da Conceicao (Other); Instituto de Infectologia Emílio Ribas (Unknown)
Responsible Party: Principal Investigator, Raquel Malaguthi de Souza, Beatriz Grinsztejn, MD, PhD, Evandro Chagas National Institute of Infectious Disease
Other Study IDs: 32449420.4.1001.5262
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Hospitalization
Keywords: Covid-19; hospitalization; biomarkers
MeSH Terms: conditions — COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total participants: 3500 participants that will have their medical forms checked
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Clinical and sociodemographic data collected through interview at admission and results of complementary tests performed during hospitalization.

SUMMARY:
The RECOVER SUS-BRASIL network, made up of excellent academic and research institutions, was formed in response to the emergence of unprecedented public health related to SARS-CoV-2. The Network's objectives are the production of scientific knowledge, the technical and scientific strengthening of participating centers, the sharing of information and experiences with other assistance services and the generation of evidence for public health policies in Brazil. The present proposal aims to increase the magnitude of the Network, proposing two studies to assess the epidemic of COVID-19 in Brazil. The first study deals with the establishment of a prospective cohort of patients hospitalized for COVID-19. Through using standardized data collection procedures, biological samples and biomarkers, this study will be able to describe clinical presentation, severity, risk factors for worsening of the disease. Multiple clinical outcomes of severity of disease, organ dysfunction, hospital mortality, length of hospital stay, hospital readmission and early post-discharge death. Will be biomarkers of inflammation, cellular and humoral immunity were also evaluated to study their association with clinical outcomes, variability of SARS-CoV-2 and the development of immunity in infected individuals through the detection and titration of neutralizing antibodies anti-SARS-CoV-2. The second study 2 will evaluate the COVID-19 epidemic in people living with HIV / AIDS, using SUS databases, such as SIM, SICLOM and SISCEL. This study is particularly relevant since on the one hand it includes a population potentially at greater risk of developing severe forms of the disease, given their underlying condition, as, on the other hand, they are exposed chronically to drugs that could potentially have an effect on SARS-CoV-2. Finally, a major objective of RECOVER SUS-BRASIL is integrate technical and scientific capacities generating scientific production of high relevance and impact and strengthening health and science throughout the country.

DETAILED DESCRIPTION:
Study 1 procedures are clinical and sociodemographic data collected through interview at admission and results of complementary exams performed during hospitalization. Data will be collected during the participant's inclusion visit (Day 0,equivalent to the date of hospital admission) and subsequently according to in-hospital visits untill discharge moment.

The team of researchers will have access to the electronic medical record or, as the case, to the paper medical record for the collection of data and variables of the study interest, and questionnaires with specific questions from participants or family members.

A visit in 31-60 days will be made, by telephone contact, for the application by a health professional of a questionnaire on mental health and verification of the occurrence of death or hospital readmission. The mental health questionnaire includes tracking disorders, such as: depression, anxiety, post-traumatic stress disorder, suicidal ideation and insomnia [questionnaires PHQ-9, GAD-7, Abbreviated PCL-C and Index Severity of Insomnia], in addition to a questionnaire on social support [MSPSS]. Patients identified with health disorders over the telephone will be referred to specialized care by a psychiatrist. Study 2 - Data from information systems drug dispensation (SICLOM - http://www.aids.gov.br/pt-br/gestores/sistemas-de-informacao/sistema-de-controle-logistico-demedicamentos-siclom), laboratory tests (SISCEL - http : //www.aids.gov.br/pt-br/sistema-de-informacao/sistema-de-controle-de-exameslaboratoriais-da-rede-nacional-de-contagem-de), information on mortality (SIM - http://sim.saude.gov.br/) and COVID-19 case notification database will be released to the Ministry of Health, with data identified with patient name, mother's name and date of birth to enable the linkage process. This sensitive data is obtained through specific forms, which include confidentiality clauses of the data. All transport and storage of this data, whether by digital physical means (for example, CD) or via the web, will be done in encrypted form with a strong algorithm. The final database will be de-identified to guarantee the confidentiality of the participants.

ELIGIBILITY:
Inclusion Criteria:Adults aged 18 years. Hospitalized for suspicious signs and symptoms of COVID-19 infection by the medical care team or confirmed by laboratory tests such as RT-PCR or rapid tests.

Exclusion Criteria:Patient or family member refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years. Hospitalized for suspicious signs and symptoms of COVID-19 infection by the medical care team or confirmed by laboratory tests such as RT-PCR or rapid tests.
Sampling Method: Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-10-25 (Estimated); Study Completion 2022-03-25 (Estimated)

PRIMARY OUTCOMES:
The main outcome of the study is hospital mortality | 25/05/2021

SECONDARY OUTCOMES:
Length of hospital stay | 25/05/2021

CONTACTS AND LOCATIONS:
Locations (13):
- Brazil (13):
  - Hospital São José de Doenças Infecciosas - HSJ / Secretaria de Saúde Fortaleza, Fortaleza, Ceará
  - Hospital Couto Maia/SES/BA, Salvador, Estado de Bahia
  - Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital dos Servidores do Estado/RJ, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Gaffree e Guinle/HUGG/UNIRIO, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Pedro Ernesto/UERJ, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional de Infectologia Evandro Chagas (Fiocruz), Rio de Janeiro, Rio de Janeiro
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Santa Maria/ Pró-Reitoria de PósGraduação e Pesquisa, Santa Maria, Rio Grande do Sul
  - Hospital Regional de São José, São José, Santa Catarina
  - Hospital Estadual Sumaré Dr. Leandro Francheschini, Sumaré, São Paulo
  - Instituto de Infectologia Emílio Ribas, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided